CLINICAL TRIAL: NCT01042405
Title: Development of a Risk Computerized Predictive Method in HD Patients by Nutritional Scoring & Assesment of NIR Method for Cr Determination
Brief Title: Nutrition Based Computerized Predictive Method for Morbidity & Mortality Risk in HD Patients. Assisng NIR for Blood Cr
Acronym: Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Zvi Barnea, Senior Nephrologist, Wolfson Medical Center
Other Study IDs: 0074-09-WOMC
Record Dates: First submitted 2010-01-01; First posted 2010-01-05 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition; Inflammation; Morbidity; Mortality
MeSH Terms: conditions — Malnutrition; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The samples were kept for additional NIR determination of Cr
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to develop a simple computer program, evaluating nutritional status of HD patients. The programming will enable to perform a nutritional screening, based on biochemical measures, taken as part of HD patients' routine care every month. The program will identify patients at risk of malnutrition, define the degree of malnutrition, and identify patients who at risk for increased morbidity and mortality. Patients who are at risk of malnutrition will be treated by a standard nutrition; dietary counseling (high protein diet, appropriate calories intake and use of oral supplementation. Intra-dialytic parenteral nutrition (IDPN) will be used for patients who fail to improve nutrition status by standard nutrition care, as a second line treatment. The effect of IDPN on their nutrition status will be evaluated. A sub group of 30 patients will provide blood smample to assess a NIR method for Cr determination as creatinine is one of the parameters our nutrition score is based on.

DETAILED DESCRIPTION:
30 patients will randomly be selected for SGA examination and comparison to the MARK results every month. Frequency and duration of hospitalizations within the 5-month collection period will documented, mortality will be documented as well. Effect of different nutritional supplementations or IDPN will be assessed. The MARK nutrition screening will be used for all patients at the beginning of every month. Monthly Biochemical data using a blood sample taken immediately before dialysis will be used to calculate a value between 0-100 showing patient's monthly nutritional status. Data for the SGA will be collected for the same dialysis patients randomly selected at the same month. The nutritional state of the patients according to the SGA will be assessed by two investigators. A statistical test will be held for agreement between observers (Cohen's k concordant coefficient).

A sub group of 30 patients will provide blood smample to assess a Near Infra Red (NIR) method for Cr determination. Application of chemometric approach will serve for constructing a fitting curve between tradtional CR measurment with NIR method.

ELIGIBILITY:
Inclusion Criteria:

* All dialysis patients in Wolfson Medical Center dialysis unit above the age of 18 years and on dialysis more than 3 months.

Exclusion Criteria:

* Patients with bilateral plegia. Hemiplegic organs of a patient (not the entire patient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients on hemodialysis, Wolfson Hospital
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2010-02 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel